CLINICAL TRIAL: NCT02273869
Title: The Influence of Rheumatologic Diseases on Fertility and Ovarian Reserve
Brief Title: Assessment of Ovarian Reserve in Women With Rheumatologic Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC-011413-CTIL
Record Dates: First submitted 2014-09-29; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatologic Diseases; Ovarian Reserve; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum blood test
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Our infertility unit has started a clinic for women with rheumatological diseases. those women are prone to infertility problems and it might be due to their illness or cytotoxic treatment . In our study we are going to observe the effect of their disease on ovarian reserve. we will assess it by using intravaginal sonography and blood test such as hormonal profile and anti-mullerian hormone (AMH).

ELIGIBILITY:
Inclusion Criteria:

* Rheumatologic disease

Exclusion Criteria:

* none

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women in reproductive age with rheumatoligic disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
hormone profile | 4 years
  Assessment of ovarian function using hormone profile and AMH levels in serum, in women with rheumatologic disease.
antral follicular count | 4 years
  we will use sonography to assess the antral follicular count as a parameter for ovarian reserve in women with rheumatologic disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Sapir Medical Center, Meir Hospital, Kfar Saba, Israel, Israel